CLINICAL TRIAL: NCT03554213
Title: Evaluation of a Typhoid Conjugate Vaccine Introduction Program in Navi Mumbai, India
Brief Title: Typhoid Conjugate Vaccine Introduction in Navi Mumbai, India
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); World Health Organization (Other); National Institute of Cholera and Enteric Diseases, India (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Stephen P Luby, Professor, Stanford University
Other Study IDs: IRB-39627; OPP1169264 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2018-05-30; First posted 2018-06-13 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Enteric Fever; Typhoid Fever; Salmonella Typhi Infection
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * In the hospital surveillance component, blood cultures will be collected and tested for Salmonella Typhi and Paratyphi. Purified bacterial isolates of Salmonella Typhi and Paratyphi will be tested for antimicrobial resistance and stored for possible future genetic/genomic testing of the bacterial DNA.
  * In a subset of the community surveillance component, dried blood spots will be collected onto filter paper and stored to test for antibodies against typhoid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1: TCV in 2018: Children receiving TCV (typhoid conjugate vaccine) in 2018 vaccination campaign by NMMC.
  Interventions: Biological: Typhoid Conjugate Vaccine
- Phase 2: TCV in 2019: Children receiving TCV (typhoid conjugate vaccine) in 2019 vaccination campaign by NMMC.
  Interventions: Biological: Typhoid Conjugate Vaccine

INTERVENTIONS:
Biological: Typhoid Conjugate Vaccine — Typbar TCV Vi-TT (Vi capsular polysaccharide conjugated with tetanus toxoid protein) manufactured by Bharat Biotech International Limited

SUMMARY:
The purpose of this study is to evaluate the impact of a government-led typhoid conjugate vaccine introduction program on typhoid disease burden in Navi Mumbai, India.

DETAILED DESCRIPTION:
A new generation of typhoid conjugate vaccines (TCVs) have been shown to be safe and provide long-lasting immunity in children. In India, Typbar TCV Vi-TT (Vi capsular polysaccharide conjugated with tetanus toxoid protein) is manufactured by Bharat Biotech International Limited (BBIL). Immunogenicity studies by BBIL showed >90% detectable antibodies to Typbar TCV vaccine at 42 days and >70% at 720 days in persons 2-45 years old. A single dose of vaccine was effective in children 6-23 months old with 98% seroconversion at 42 days and persistent high antibody titers at 720 days. Another randomized controlled trial study by University of Oxford tested Vi-TT with a human challenge model of typhoid fever in which participants ingested Salmonella Typhi after vaccination. Typhoid fever was diagnosed by clinical criteria and/or positive blood culture at 2 weeks in 77% of controls (n=31) as compared to 35% in the Vi-TT group (n=37) to give vaccine efficacy of 54% (95% confidence interval of 26-71). Typbar TCV has been licensed in India for children >6 months old since 2013 and is currently used in the private sector. In January 2018, the World Health Organization (WHO) recommended the use of typhoid conjugate vaccines especially in those countries with the highest burden of disease and the highest burden of antimicrobial resistance. However, there are no field effectiveness studies yet for Typbar TCV.

In this study, a hybrid facility- and community-based typhoid surveillance strategy will be used to evaluate the impact of a government-led typhoid conjugate vaccine introduction program on typhoid disease burden in Navi Mumbai, India. Navi Mumbai is a metropolitan area extending from Mumbai with approximately 1.4 million people and wide demographic and socioeconomic strata, including slums. Navi Mumbai is comprised of 13 area nodes, and 8 of these nodes are under the jurisdiction of the local government body, Navi Mumbai Municipal Corporation (NMMC). Navi Mumbai has high enteric fever burden: a 2008 study found 98 blood culture-confirmed pediatric cases over 16 months in 2 hospitals with a majority of isolates exhibiting multi-drug resistance. Data from one private laboratory in 2015 showed over 225 S. Typhi cases including 3 cases with ceftriaxone resistance.

NMMC has decided to introduce TCV into public sector routine immunization services and will vaccinate all children 9 months to <15 years old within its jurisdiction - estimated 390,000 children - with TCV over 2 years. NMMC government officials are collaborating with researchers from WHO India, Institute of Cholera and Enteric Diseases (NICED), Centers for Disease Control and Prevention (CDC), and Stanford University to implement the TCV introduction in a two-phase cluster-randomized program in order to allow rigorous evaluation of population impact. NMMC has 22 urban health posts (UHPs) that give routine childhood immunizations. UHPs were first grouped into 3 strata based on % of population living in slums: low, medium, or high. Half of the UHPs within each stratum were then randomly selected to receive TCV in 2018 (Phase 1) and the remaining UHPs to receive TCV one year later in 2019 (Phase 2).

Evaluation studies of NMMC's TCV introduction program include: impact on blood-culture confirmed typhoid fever; impact on clinical syndromes of febrile illness; vaccine safety; vaccine efficacy; vaccination campaign coverage and acceptability surveys; environmental water contamination with Salmonella Typhi; seroconversion associated with typhoid infection; and cost-effectiveness of typhoid conjugate vaccination campaign.

ELIGIBILITY:
Inclusion Criteria:

For overall study,

1. For hospital-based surveillance, children age 6 months to 16 years.
2. For community-based surveys, adult members of households with children <16 years old.
3. Parental consent (and child assent for >12 years) given.

For hospital-based surveillance for typhoid fever, additional criteria include: history of fever for >72 hours within the last 7 days without upper respiratory tract symptoms and vesicular rash; strong clinical suspicion of enteric fever including ileal perforations; or diagnosis of enteric fever confirmed by positive blood cultures or histopathology. For outpatients, additional criterion of living in areas governed by Navi Mumbai Municipal Corporation.

For hospital-based surveillance of adverse events of special interest, timing will focus on one month prior to and 42 days after the vaccination campaign. Diagnoses included are: anaphylaxis, bronchospasm, urticaria, Guillain-Barré syndrome, meningitis, encephalitis, myelitis, seizures, thrombocytopenia, and sudden death.

For all community surveys, additional criterion of living in areas governed by Navi Mumbai Municipal Corporation.

Exclusion Criteria:

For all study components,

1. Already enrolled in same study component.
2. No informed consent or assent given.

For hospital-based surveillance for typhoid fever, additional exclusion criteria are: fever <72 hours, symptoms of upper respiratory tract infection (coryza, rhinorrhea), and vesicular exanthem. For outpatients, those living outside of NMMC-governed areas will be excluded.

For community surveys, households without children <16 years old and households in which there is no adult (>18 years old) at time of survey will be excluded.

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The focus of this study is children age 6 months to 16 years living in areas governed by Navi Mumbai Municipal Corporation (NMMC). The age range of children eligible to receive typhoid conjugate vaccine (TCV) in NMMC's TCV introduction program is 9 months to 15 years. For community surveys, only households with children <16 years old will be selected.
  The evaluation study will examine a slightly broader age range than NMMC's TCV vaccination program because TCV is licensed for >6 month old children and because the vaccine introduction will occur over 1 year thus the oldest eligible children will be 16 years old at study end.
Sampling Method: Probability Sample
Enrollment: 17292 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
blood culture-confirmed typhoid fever | up to 24 months
  Hospital surveillance for typhoid fever diagnosed by blood cultures will be conducted at 6 study sites in Navi Mumbai: 5 hospitals and 1 independent laboratory.

SECONDARY OUTCOMES:
Adverse events following immunization | up to 4 months
  Evaluation of safety and adverse events following immunization (AEFI) during Phase I of TCV introduction in 2018. Three safety evaluations include: 1) routine national AEFI surveillance system reports, 2) active follow-up by phone of a subset of vaccine recipients at 48hrs and 7 days post vaccination, and 3) hospital-based surveillance at 5 hospital study sites conducting typhoid fever surveillance examining patient records for adverse events of special interest in both vaccinated and unvaccinated populations
vaccination coverage | up to 18 months
  Community surveys estimating TCV coverage achieved by the vaccination campaign in the public sector during phase 1 (and potentially phase 2 if funding allows) as well as vaccine acceptability, refusals, knowledge, attitudes, and social mobilization strategies.
environmental water contamination with Salmonella Typhi | up to 24 months
  Molecular testing of household and municipal water samples for presence of Salmonella Typhi and Paratyphi A and impact of TCV vaccination program on water contamination.
seroconversion associated with typhoid infection | up to 24 months
  Collect dried blood spots in subset of household surveys and store for future testing of antibodies associated with typhoid infection (once other research studies on best antibody tests have resulted).
cost-effectiveness of typhoid conjugate vaccination campaign | up to 24 months
  Plan to develop a tool and to estimate the delivery cost of TCV, to estimate the cost of illness (COI) related to typhoid fever, and ultimately to estimate the cost-effectiveness of typhoid conjugate vaccination campaign conducted in Navi Mumbai.
clinical syndromes of febrile illness | up to 18 months
  Community-based surveys of clinical syndromes of febrile illness and healthcare utilization in NMMC-governed areas (same as TCV vaccination areas).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Luby, MD, Principal Investigator — Stanford University; Kashmira Date, MD MPH, Principal Investigator — Centers for Disease Control and Prevention; Shanta Dutta, MD PhD, Principal Investigator — National Institute of Cholera and Enteric Diseases (NICED); Pankaj Bhatnagar, MD, Principal Investigator — World Health Organization (WHO) - India
Locations (6):
- India (6):
  - D. Y. Patil Medical College and Hospital, Nerul, Navi Mumbai
  - Dr. Joshi's Central Clinical Microbiology Laboratory, Vashi, Navi Mumbai
  - Dr. Yewale Multispecialty Hospital for Children, Vashi, Navi Mumbai
  - Mahatma Gandhi Memorial (MGM) New Bombay Hospital, Vashi, Navi Mumbai
  - Mathadi Hospital Trust, Koparkharaine, Navi Mumbai
  - Navi Mumbai Municipal Corporation (NMMC) General Hospital, First Referral Unit (FRU), Vashi, Navi Mumbai